CLINICAL TRIAL: NCT00810927
Title: Role of NO in the Control of Choroidal Blood Flow During a Decrease in Ocular Perfusion Pressure
Brief Title: Role of Nitrogen Oxide (NO) in the Control of Choroidal Blood Flow During a Decrease in Ocular Perfusion Pressure
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Gabriele Fuchsjaeger-Mayrl, MD, Department of Clinical Pharmacology, Medical University of Vienna
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: OPHT-270602
Record Dates: First submitted 2008-12-17; First posted 2008-12-18 (Estimated); Last update posted 2008-12-18 (Estimated); Status verified 2008-12

CONDITIONS: Physiology, Ocular; Microcirculation; Regional Blood Flow; Autoregulation
MeSH Terms: interventions — Laser-Doppler Flowmetry

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Active Comparator): Phenylephrine (Neosynephrine®, Abbott Laboratories, North Chicago, IL, USA) dose: 1µg/(kg.min), infusion period 20 minutes
  Interventions: Procedure: Suction cup application; Procedure: Laser Doppler flowmetry; Procedure: Measurement of intraocular pressure
- 2 (Active Comparator): NG-monomethyl-L-arginine (L-NMMA, Clinalfa, Läufelfingen, Switzerland) dose: bolus 6mg/kg over 5 minutes followed by a continuous infusion of 60µg/(kg.min) over 15 minutes
  Interventions: Procedure: Suction cup application; Procedure: Laser Doppler flowmetry; Procedure: Measurement of intraocular pressure
- 3 (Placebo Comparator): Physiologic saline solution
  Interventions: Procedure: Suction cup application; Procedure: Laser Doppler flowmetry; Procedure: Measurement of intraocular pressure

INTERVENTIONS:
Procedure: Suction cup application — he IOP will be raised by a 11 mm diameter, standardized suction cup placed on the temporal sclera with the anterior edge at least 1 mm from the limbus.
Procedure: Laser Doppler flowmetry — Measurement of choroidal blood flow
Procedure: Measurement of intraocular pressure

SUMMARY:
Autoregulation is the ability of a vascular bed to maintain blood flow despite changes in perfusion pressure. For a long time it had been assumed that the choroid is a strictly passive vascular bed, which shows no autoregulation. However, recently several groups have identified some autoregulatory capacity of the human choroid. In the brain and the retina the mechanism behind autoregulation is most likely linked to changes in transmural pressure. In this model arterioles change their vascular tone depending on the pressure inside the vessel and outside the vessel. In the choroid, several observations argue against a direct involvement of arterioles. However, the mechanism behind choroidal autoregulation remains unclear.

In the present study autoregulation of the choroid will be investigated during a decrease in ocular perfusion pressure, which will be achieved by an increase in intraocular pressure. Pressure/flow relationships will be investigated in the absence or presence of a NO synthase inhibitor. As a control substance the alpha-receptor agonist phenylephrine will be used.

ELIGIBILITY:
Inclusion Criteria:

* Men aged between 19 and 35 years, nonsmokers
* Body mass index between 15th and 85th percentile (Must et al. 1991)
* Normal findings in the medical history and physical examination unless the investigator considers an abnormality to be clinically irrelevant
* Normal laboratory values unless the investigator considers an abnormality to be clinically irrelevant
* Normal ophthalmic findings, ametropia < 3 Dpt.

Exclusion Criteria:

* Regular use of medication, abuse of alcoholic beverages, participation in a clinical trial in the 3 weeks preceding the study
* Treatment in the previous 3 weeks with any drug
* Symptoms of a clinically relevant illness in the 3 weeks before the first study day
* History of hypersensitivity to the trial drug or to drugs with a similar chemical structure
* History or presence of gastrointestinal, liver or kidney disease, or other conditions known to interfere with, distribution, metabolism or excretion of study drugs
* Blood donation during the previous 3 weeks

Ages: 19 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2003-09; Primary Completion 2004-02 (Actual); Study Completion 2005-08 (Actual)

PRIMARY OUTCOMES:
ocular perfusion pressure - choroidal blood flow relationship

CONTACTS AND LOCATIONS:
Overall Officials: Gabriele Fuchsjäger-Mayrl, MD, Principal Investigator — Department of Clinical Pharmacology, Medical University of Vienna
Locations (1):
- Department of Clinical Pharmacology, Medical University of Vienna, Vienna, Austria